CLINICAL TRIAL: NCT02435810
Title: Natural History Study of Inflammatory and Infectious Diseases of the Nervous System
Brief Title: Inflammatory and Infectious Diseases of the Nervous System
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150125; 15-N-0125
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12-30

CONDITIONS: Brain Disease
Keywords: Neuroinflammation; Infections; Natural History
MeSH Terms: conditions — Brain Diseases; Neuroinflammatory Diseases; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family Member: A family member of a patient with known or suspected infection or inflammation of the nervous system based on clinical or imaging data provided
- Patient: Patient with known or suspected infection or inflammation of the nervous system based on clinical or imaging data provided

SUMMARY:
Background:

- Inflammation is how the body reacts to infection or injury. Infections or inflammation in the brain and nerves can be serious. There aren t always good tests to detect this. Researchers want to learn more about how diseases affect the brain and nerves to develop better tests and treatments.

Objective:

- To learn more about how inflammation and infections hurt the brain and nervous system.

Eligibility:

- People at least 2 years old with a diagnosis or suspected diagnosis of nervous system infection or inflammation.

Design:

* For some participants, a clinician outside of NIH will collect blood, tissue, and other samples. These will be sent to NIH and analyzed.
* Other participants will have several visits to NIH. Children may not have all these tests.
* Participants will have:
* Medical history.
* Physical and neurological exam.
* Blood and urine samples collected.
* Saliva collected. They will chew on a piece of sterile cotton for one minute.
* Magnetic resonance imaging (MRI) scan. The scanner is a metal cylinder in a strong magnetic field. Participants will lie on a table that slides in and out of the cylinder. Participants will get a contrast agent through an intravenous (IV) catheter during the MRI. A needle will be used to guide a thin plastic tube (catheter) into an arm vein.
* Lumbar puncture. Skin will be numbed and a needle will be inserted into the space between the bones in the back. Fluid will be removed.
* Some participants may have optional study procedures. These may include eye tests, memory and thinking testing, tests with electrodes on the head, or skin biopsy.

DETAILED DESCRIPTION:
Objective:

The objective of this study is to examine the natural course of infectious and inflammatory diseases of the nervous system, to identify causative or associated pathogens when unknown, and generally to better understand the underlying immunological, genetic and pathophysiologic mechanisms that cause and contribute to these diseases and their ultimate neurological outcomes.

Study Population:

The study population will be patients at least 2 years old with known or suspected infection or inflammation of the nervous system and family members. Participants will be recruited through referrals to the NIH.

Design:

This is a longitudinal case series with standardized research data collection at predefined time points. Participants will have scheduled visits at the NIH either as an outpatient or an inpatient. The core research evaluations include: a comprehensive history and neurological examination; blood collection; neuroimaging; and lumbar puncture. Follow up visits will be individualized based on clinical needs and results of research evaluations. For some participants, no additional NIH visits will be necessary.

Additionally, we will also enroll participants with known or suspected infections or inflammation of the nervous system from whom only biological samples collected by outside clinicians will be processed and retained for research analyses. In cases were samples remain from those collected for clinical reasons and the samples are deidentified, the samples may be obtained with a waiver of informed consent.

Outcome Measures:

The study outcomes will primarily be the characterizations of varied inflammatory and infectious nervous system diseases. These characterizations will include: the clinical phenotype and biomarkers.

ELIGIBILITY:
* INCLUSION CRITERIA:

At the time of enrollment, participants will:

1. Have a known or suspected infection or inflammation of the nervous system or post infection sequelae based on clinical or imaging data provided by the referral facility. For the purpose of this study, neuroinfectious disease or neuroinflammation is defined as any of the following:

   1. fever with nervous system signs or symptoms (excluding delirium)
   2. any neurological symptoms accompanied by cerebrospinal fluid (CSF) with evidence of inflammation (which may include pleocytosis, hypoglycorrachia, elevated protein, or other evidence of intrathecal immune activation including IgG index or presence of oligoclonal bands)
   3. systemic infection or inflammatory disease with neurological involvement
   4. neuroimaging suggestive of infection or inflammation (for example, presence of contrast-enhancing lesions on CT or MRI)
   5. clinical presentation suggestive of infection or inflammatory process of the nervous system without better explanation
   6. history of infection or inflammatory process of the nervous system
2. Be willing to participate in the protocol s procedures, unless clinically contraindicated
3. Be willing to provide informed consent, either directly or via appointed legally authorized representative
4. Be willing to consent for collection of clinical data or biological samples or their cryopreservation
5. Be at least 2 years old

INCLUSION CRITERIA FOR PROCESSING OF BIOLOGICAL SAMPLES ONLY:

At the time of enrollment, participants will:

1. Have a known or suspected infection or inflammation of the nervous system or post infection sequelae based on clinical or imaging data provided by the referral facility. For the purpose of this study, neuroinfectious disease or neuroinflammation is defined as any of the following:

   1. fever with nervous system signs or symptoms (excluding delirium)
   2. any neurological symptoms accompanied by cerebrospinal fluid (CSF) with evidence of inflammation (which may include pleocytosis, hypoglycorrachia, elevated protein, or other evidence of intrathecal immune activation including IgG index or presence of oligoclonal bands)
   3. systemic infection or inflammatory disease with neurological involvement
   4. neuroimaging suggestive of infection or inflammation (for example, presence of contrast-enhancing lesions on CT or MRI)
   5. clinical presentation suggestive of infection or inflammatory process of the nervous system without better explanation
   6. history of infection or inflammatory process of nervous system
2. Be willing to provide informed consent, either directly or via appointed legally authorized representative
3. Be willing to consent for collection of clinical data or biological samples or their cryopreservation
4. Be at least 2 years old

EXCLUSION CRITERIA:

At the time of enrollment, participants will:

1. Not have a clinically significant medical condition that, in the best judgment of the investigators, may expose the patient to undue risk of harm or prevent the patient from completing the study (examples include, but are not limited to, ischemic cardiomyopathy, clotting disorder, brittle diabetes)
2. Not have an acute or unstable medical condition that, in the best judgement of the investigator, would be difficult to handle at the NIH Clinical Center
3. Not have a clearly-established diagnosis of well-characterized disease entity with validated treatment algorithms for which proposed resource investment, in the opinion of the investigators, would not contribute to further advancement of knowledge

EXCLUSION CRITERIA FOR PROCESSING OF BIOLOGICAL SAMPLES ONLY:

At the time of enrollment, participants will not have:

1. A clearly-established diagnosis of well-characterized disease entity with validated treatment algorithms for which proposed resource investment, in the opinion of the investigators, would not contribute to further advancement of knowledge

INCLUSION CRITERIA FOR FAMILY MEMBERS:

1. Have a family member enrolled on 15-N-0125
2. Be at least 2 years old
3. Be able to provide informed consent and comply with study procedures

EXCLUSION CRITERIA FOR FAMILY MEMBERS:

1. Not willing to consent for collection of biological samples or their cryopreservation

Ages: 2 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will have a known or suspected infection or inflammation of the nervous system based on clinical or imaging data provided.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-05-06 (Actual); Primary Completion 2026-11-29 (Estimated); Study Completion 2026-11-29 (Estimated)

PRIMARY OUTCOMES:
This is a natural history study of individual cases | 12 months after the last participant is enrolled.
  To describe the natural history of inflammatory and infectious diseases of the nervous system and to investigate the relative contribution of underlying pathophysiological processes to morbidity, response to treatment and outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Avindra Nath, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-N-0125.html